CLINICAL TRIAL: NCT04167709
Title: Child Health Services Nurses Clinical Competence in Detecting Signs of Post Partum Depression in Non-Native-Speaking Immigrant Mothers' -Development, Testing and Evaluation of an Intervention
Brief Title: CHS Nurses Clinical Competence in Detecting Signs of PPD in Non-Native Speaking Immigrant Mothers'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other); Föreningen Mjölkdroppen Helsingborg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018/1063
Record Dates: First submitted 2019-11-04; First posted 2019-11-19 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Depression, Postpartum
Keywords: postpartum depression; immigrant women; Child Health Services; nurse; Edinburgh Postnatal Depression Scale
MeSH Terms: conditions — Depression, Postpartum | interventions — Educational Status; Clinical Competence

STUDY DESIGN:
Intervention Model Description: The study has a pre-post experimental design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allocated CHS nurses (Experimental): Primary and secondary baseline data are collected from the allocated CHS nurses before the study starts. The CHS nurses are then given the educational intervention and afterwards primary and secondary outcomes are collected again.
  Interventions: Other: Education in clinical competence in detecting signs of postpartum depression in immigrant mothers

INTERVENTIONS:
Other: Education in clinical competence in detecting signs of postpartum depression in immigrant mothers — Groupbased educational intervention aimed at nurses in the Child Health Services in strengthening clinical competence in detecting signs of postpartum depression in non-native-speaking immigrant mothers

SUMMARY:
The aim is to develop, test and evaluate an educational intervention with the purpose to strengthen Child Health Services (CHS) Nurses clinical competence in detecting signs of postpartum depression in non-native-speaking immigrant mothers. The pilot study has a pre-post experimental design. Data are collected before and after the intervention. The differences in the values of the collected data are used to estimate the effect of the intervention.

DETAILED DESCRIPTION:
To be eligible for the study the CHS nurse must perform screening of immigrant mothers for postpartum depression with help of an interpreter according to the Edinburgh Postnatal Depression Scale (EPDS) method more than three times a year. The EPDS is a likert form scale with ten statements and is used in combination with a Clinical interview.

Approximately 40-45 CHS nurses will be enrolled in the pilot study. The number of nurses are calculated in comparison to two other published studies within the same context. The instruments Clinical Cultural Competence Training Questionnaire (CCCTQ) and General Self-Efficacy scale (GSE) will be used as primary outcomes measures. Data are collected before the first education day and after the second education day. Secondary outcomes are also collected in connection to the educational intervention and consists of reported yearly statistics; how many mothers were are offered screening, participated in screening, number of screenings preformed with help og an interpreter and number of mothers offered follow-up after participating in screening.

ELIGIBILITY:
Inclusion Criteria:

* Nurse specialized in Primary Healthcare Nursing or Pediatric Nursing
* Employed in the Child Health Services in the County Scania in Sweden
* Performing at minimum three screenings per year for postpartum depression, according to the EPDS-method, with help of an interpreter

Exclusion Criteria:

-

Ages: 25 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-09 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical Cultural Competence Training Questionnaire | the questionnaire are given before and directly after the educational intervention
  measures change in the participants experienced cultural competence. Consist of 8 items. Responses are made on a 4-pointscale.The mean score is calculated by adding up the sum of all answers (range 8-32) and dividing it by 8. The higher score the better outcome.
General Self Efficacy scale | the questionnaire are given before and directly after the educational intervention
  measures change in the participants confidence in their own ability. Consist of 10 items. Responses are made on a 4-pointscale.The mean score is calculated by adding up the sum of all answers (range 10-40) and dividing it by 10. The higher score the better outcome.

SECONDARY OUTCOMES:
mothers offered to participate in screening | before the educational intervention are given and one year after the educational intervention are given
  number of mothers offered to participate in screening for postpartum depression
mothers participating in screening | before the educational intervention are given and one year after the educational intervention are given
  number of mothers participating in screening for postpartum depression
screening with help of interpreter | before the educational intervention are given and one year after the educational intervention are given
  number of screenings performed with help of an interpreter
mothers offered follow-up after screening | before the educational intervention are given and one year after the educational intervention are given
  number of mothers offered follow-up after participating in screening for postpartum depression

CONTACTS AND LOCATIONS:
Overall Officials: Inger Kristensson Hallström, professor, Study Chair — Lund University, Faculty of Medicine, Department of Health Sciences
Locations (1):
- Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
Since this is a small pilot study a study protocol will not be published.

REFERENCES:
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Result] Love J, Moore CD, Hensing G. Validation of the Swedish translation of the General Self-Efficacy scale. Qual Life Res. 2012 Sep;21(7):1249-53. doi: 10.1007/s11136-011-0030-5. Epub 2011 Oct 8. PMID 21984467
- [Derived] Skoog M, Rubertsson C, Kristensson Hallstrom I. Feasibility of an evidence-based educational intervention in screening immigrant mothers for postpartum depression: A pretest-posttest experimental design. Scand J Caring Sci. 2023 Mar;37(1):173-184. doi: 10.1111/scs.13086. Epub 2022 May 6. PMID 35524434
- See also: European Community contract no. 2013 62 09 — https://www.mem-tp.org/pluginfile.php/1161/mod_resource/content/1/2013%2062%2009_MEM_TP%20Interim%20Report_March_2015.pdf
- See also: Medical Research Councils framework for complex interventions — http://www.mrc.ac.uk/index.cfm/searchresults/?keywords=complex+interventions&display=search&newSearch=true&noCache=1